CLINICAL TRIAL: NCT06096948
Title: Safety and Efficacy of a New Hemostatic System to Prevent Delayed Bleeding After Endoscopic Resection in a Selected High-risk Population
Brief Title: Nexpowder to Prevent Delayed Bleeding After Endoscopic Resection
Acronym: NEX-ENDOHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Lemmers Arnaud, Professor Endoscopy Unit, Director of Clinic Department of Gastroenterology, Hepatopancreatology and Digestive Oncology Erasme Hospital,, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NEXPOWDER-ENDOHS; P2023/250 (Other: ERASME ETHICS COMMITTEE); B4062023000141 (Other: ERASME ETHICS COMMITTEE)
Record Dates: First submitted 2023-10-10; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Gastro Intestinal Bleeding; Polyps
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NEXPOWDER-ENDOHS (Experimental): Standard of care ESD or EMR procedure and application of Nexpowder on the resection site to prevent delayed bleeding.
  Interventions: Device: NEXPOWDER-ENDOHS

INTERVENTIONS:
Device: NEXPOWDER-ENDOHS — Standard of care ESD or EMR procedure and application of Nexpowder on the resection site to prevent delayed bleeding.

SUMMARY:
Safety and effectiveness of a new hemostatic system to prevent delayed bleeding after endoscopic resection in a selected high-risk population (NEXPOWDER- ENDOHS).

Indication:

Patients with indication of endoscopy resection by endoscopic mucal resection (EMR) or endoscopic submucosal dissection (ESD) with high risk of delayed bleeding (≥5%).

Hypotheses:

The use of NexpowderTM after upper and lower gastrointestinal ESD or EMR of ≥20mm in high-risk population will prevent and decrease delayed bleeding to less than 5%.

DETAILED DESCRIPTION:
Hypotheses:

The use of NexpowderTM after upper and lower gastrointestinal ESD or EMR of ≥20mm in high-risk population will prevent and decrease delayed bleeding to less than 5%.

Study design:

This is an investigator-initiated, multicentric, international, open-label, non-controlled, prospective study:

* All subjects with indications undergo screening and baseline visit,
* Informed consent is obtained when scheduling the ESD or EMR procedure,
* ESD or EMR is performed, at the end of resection, NexpowderTM is applied on the resected field,
* A follow up visit is scheduled at 4 weeks.

Endpoints:

* Primary:
* Assess the delayed bleeding rate after ESD or EMR of ≥20mm in a selected high-risk population when using NexpowderTM at the end of the procedure.

This hypothesis is that the use of NexpowderTM will reduce the rate of DB from 16% (reported rate in the literature) to less than 5% (excepted observed rate during the study).

* Secondary:
* Safety of NexpowderTM endoscopic hemostasis system,
* Procedure duration and NexpowderTM spaying duration,
* Length of stay in hospital,
* Post intervention pain,
* Adverse events related to the use of NexpowderTM:
* Per procedural
* Early (up to controlled endoscopy or at 24hours post procedure)
* Late (up to 4 weeks follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 year of age at the time of informed consent,
* Patients must have given written informed consent,
* Subjects with documented lesions with indication of upper or lower endoscopic removal by ESD or EMR with high risk of delayed bleeding (+/-16%), namely:
* All patients under anticoagulation (vitamin K antagonist, direct anticoagulant, non-fractionated heparin or low molecular weight heparin) or anti-aggregating (P2Y12 receptor antagonists),
* Patients without anticoagulation or anti-aggregating with indication of duodenal EMR or ESD (if duodenal cold snare EMR: only under anticoagulant or P2Y12 receptor antagonist),
* Resection field of ESD or EMR is ≥ 20mm (same size restriction in case of endoscopic papillectomy).

Exclusion Criteria:

* Resection bed <20mm,
* Subject currently enrolled in another interventional confounding research (no contra-indication for image or blood collection in another protocol),
* Incapacitated subjects, pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Safety in terms of Adverse Events (AE related to Nexpowder) | 1 month
  * number of intraprocedural complications (perforation,…)
  * number of post-procedure complications (delayed perforation, peritonitis,..)
Efficacy of Nexpowder in changing the delayed bleeding rate | 1 month
  Decrease the delayed bleeding rate

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (9):
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - UZ Gasthuisberg (KUL), Leuven, Vlaams Brabant
  - AZ Sint-Jan Brugge-Oostende, Bruges, West-Vlaanderen
  - AZ Delta Campus Rumbeke, Roeselare, West-Vlaanderen
  - CHU Saint-Pierre, Brussels
  - HUB - Hôpital Erasme, Service de Gastro-Entérologie (ULB), Brussels
  - Cliniques universitaires Saint-Luc (UCL), Brussels
  - UZ Gent, Ghent
  - Groupe Santé CHC - Clinique du MontLégia, Liège
- Netherlands (3):
  - Amsterdam UMC - Location VUMC, Amsterdam
  - Amsterdam UMC - Location AMC, Amsterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No